CLINICAL TRIAL: NCT02453204
Title: STAND UP - Sedentary Behaviour in Older Adults: Investigating a New Therapeutic Paradigm Work Package 3: Investigating the Effect of Sedentary Time, Reduced Sedentary Time and Increased Light-intensity Physical Activity on Metabolic and Psychological Health in Older Adults
Brief Title: STAND UP - Sedentary Behaviour in Older Adults: Investigating a New Therapeutic Paradigm
Acronym: STAND-UP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leicester (Other)
Collaborators: University of Glasgow (Other); National Institute for Health Research, United Kingdom (Other Government); National Health Service, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 0482; MR/K025090/1 (Other Grant/Funding Number: UK Medical Research Council); CRN18120 (Registry Identifier: UK Clinical Research Network); UOLE0482 (Other: University of Leicester (Sponsor ID))
Record Dates: First submitted 2015-05-12; First posted 2015-05-25 (Estimated); Last update posted 2020-01-30 (Actual); Status verified 2016-06

CONDITIONS: Older Adults
MeSH Terms: interventions — Sitting Position; Standing Position; Walking

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Sitting (Experimental): Participants will remain sitting throughout the test period whilst undertaking typical sedentary behaviours such as watching TV, using a computer, reading and writing. Walking and standing will be restricted.
  Interventions: Behavioral: Sitting
- Standing (Experimental): Participants will be asked to break their sitting time by standing for five minutes every 30 minutes. Participants will be asked to stand in the same position with no further instructions provided. In total, individuals will accumulate 12 bouts (60 minutes) of standing throughout the test period.
  Interventions: Behavioral: Standing
- Walking (Experimental): The walking condition will be identical to standing, but the breaks in sitting time will be punctuated with five minute bouts of self-paced walking rather than standing.
  Interventions: Behavioral: Walking

INTERVENTIONS:
Behavioral: Sitting
  Arms: Sitting
Behavioral: Standing
  Arms: Standing
Behavioral: Walking
  Arms: Walking

SUMMARY:
Research has shown that reducing the time spent sitting can reduce the risk of many diseases, such as diabetes and heart disease, and improve health. It is estimated that many older adults typically spend 70% of their waking day sitting, but little is known about whether reducing sitting promotes health and well-being in this age group. The aim of this research is to investigate the health effects of reducing sitting time by replacing it with short periods of standing or walking in adults over the age of 65.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged between 65 to 79 years inclusive
* Able to walk (without any assistive devices and not requiring assistance from another person)
* Ability to communicate in and understand English to participate in the informed consent process.

Exclusion Criteria:

* Regular purposeful exercise (≥75 minutes of self-reported vigorous exercise per week)
* Inability to stand or undertake light ambulation
* Psychological condition which limits participation in the study (e.g. dementia)
* Inability to communicate or understand English
* Steroid use
* Use of glucose lowering medication
* Inability to give informed consent

Ages: 65 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 76 (Actual)
Dates: Start 2015-04; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Insulin area under the curve | 3 experimental intervention study visits over an estimated period of 1 month
  Samples will be batched and analysed at the end of the study within a certified research laboratory at the Institute of Cardiovascular and Medical Sciences (ICAMS), University of Glasgow. Samples collected at the Leicester Diabetes Centre will be sent by courier in specialist containers and packed with dry ice.

SECONDARY OUTCOMES:
Glucose area under the curve | 3 experimental intervention study visits over an estimated period of 1 month
Triglyceride area under the curve | 3 experimental intervention study visits over an estimated period of 1 month
1H NMR Metabolomics spectroscopy | 3 experimental intervention study visits over an estimated period of 1 month
  Hydrogen-1 Nuclear Magnetic Resonance assessment undertaken on blood samples collected throughout experimental intervention days
Blood pressure | 3 experimental intervention study visits over an estimated period of 1 month
Felt Arousal Scale (0-5) | 3 experimental intervention study visits over an estimated period of 1 month
  Positive affect and mood measured using the 6-point Likert Felt Arousal scale (0 = "low arousal" to 5 = "high arousal") that will be used to assess arousal.
Feeling Scale (-5 to +5) | 3 experimental intervention study visits over an estimated period of 1 month
  Positive affect and mood measured using the 11-point Likert Feeling Scale (-5 = "very bad" to +5 = "very good") will be used to assess affective valence.
Semantic Verbal Fluency Test (number of items) | 3 experimental intervention study visits over an estimated period of 1 month
  The Semantic Verbal Fluency Test assesses semantic memory and language, and participants will be asked to name as many items as they can that belong to a particular category. The categories selected for each of the experimental days will be clothing and animals.
Hopkins Verbal Learning Test (number of words recalled) | 3 experimental intervention study visits over an estimated period of 1 month
  The Hopkins Verbal Learning Test assesses verbal learning and working memory and requires immediate and delayed recall of a series of 12 words over three learning trials. Participants will be requested to undertake the delayed recall component at the end of the first set of cognitive function tests and during the second set of cognitive function tests on experimental intervention days.
Trail Making Tests A (time to complete) | 3 experimental intervention study visits over an estimated period of 1 month
  The Trail Making Tests A assesses cognitive flexibility and requires connecting randomly located numbers in numerical order (e.g. 1,2,3,4).
Trail Making Tests B (time to complete) | 3 experimental intervention study visits over an estimated period of 1 month
  The Trail Making Tests B assesses cognitive flexibility and requires connecting randomly located numbers and letters in numerical and alphabetical order alternately (e.g. 1,A,2,B,3,C).
Rapid Visual Information Processing Test (number of sequences detected and errors) | 3 experimental intervention study visits over an estimated period of 1 month
  The Rapid Visual Information Processing Test assesses sustained visual attention using numbers and requires both selective attention and working memory. This test displays a number on screen that changes between odd and even digits and individuals must detect target sequences of three odd or three even consecutive digits.
Karolinska Sleepiness Scale (1-9) | 3 experimental intervention study visits over an estimated period of 1 month
  Sleep quality measured using the 9-point Likert Karolinska Sleepiness Scale (1= "very alert" to 9= "very sleepy, fighting sleep, an effort to keep awake") based on a self-reported subjective assessment of the participant's level of drowsiness at the time.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Yates, Principal Investigator — University of Leicester
Locations (2):
- United Kingdom (2):
  - BHF Glasgow Cardiovascular Research Centre, University of Glasgow, 126 University Avenue, Glasgow
  - Leicester Diabetes Centre, Diabetes Research Unit, University of Leicester, Leicester General Hospital, Leicester

REFERENCES:
- [Derived] Yates T, Edwardson CL, Celis-Morales C, Biddle SJH, Bodicoat D, Davies MJ, Esliger D, Henson J, Kazi A, Khunti K, Sattar N, Sinclair AJ, Rowlands A, Velayudhan L, Zaccardi F, Gill JMR. Metabolic Effects of Breaking Prolonged Sitting With Standing or Light Walking in Older South Asians and White Europeans: A Randomized Acute Study. J Gerontol A Biol Sci Med Sci. 2020 Jan 1;75(1):139-146. doi: 10.1093/gerona/gly252. PMID 30403772
- See also: NIHR Leicester-Loughborough Diet, Lifestyle and Physical Activity Biomedical Research Unit — http://www.ll.dlpa.bru.nihr.ac.uk/
- See also: Leicester Diabetes Centre — http://www.leicesterdiabetescentre.org.uk/